CLINICAL TRIAL: NCT02383121
Title: Midodrine for Ischemic Stroke With Penumbra
Acronym: MISP
Status: Withdrawn | Type: Observational
Why Stopped: Changed study to an observational study
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam de Havenon, Assistant Professor, University of Utah
Other Study IDs: IRB_76683
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Midodrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No patients: Study has been withdrawn
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — Not appliciable
  Other Names: Acute ischemic patients

SUMMARY:
Acute ischemic stroke (AIS) affects over 700,000 Americans every year and is the leading cause of long-term disability. Early neurological deterioration after AIS typically occurs within 72 hours of stroke onset and affects 30% of all stroke patients, who have a higher rate of death or poor outcome. Several mechanisms account for early neurological deterioration, including hemorrhagic conversion, systemic illness, cerebral edema, and seizure, but the most common cause is extension of the stroke into the "penumbra," a region of salvageable brain tissue surrounding the core of irreversible ischemic infarct. The penumbra is tenuously perfused by collateral blood vessels. AIS management is primarily focused on recanalizing the occluded artery causing the stroke, but an alternative and relatively unexplored approach is optimization of collateral blood flow.

Over 60% of AIS patients present with a transient acute hypertensive response, which is theorized to be the result of either increased sympathoadrenal tone, poorly controlled underlying hypertension, or an unknown stroke-specific mechanism related to augmenting cerebral perfusion through collateral blood flow. Epidemiological data suggests worse stroke outcomes are associated with extremes of sustained hypo- or hypertension, which has led to dozens of clinical trials involving over 20,000 patients to determine if pharmacologically lowering blood pressure after AIS is beneficial. The results have been persistently neutral or negative. In contrast, there have been no major clinical trials on the efficacy of using vasopressor medications to maintain or increase baseline blood pressure after AIS, despite promising preclinical data and pilot studies that showed no increase in cerebral hemorrhage or edema. The only randomized trial of vasopressor use after AIS demonstrated an improvement in clinical outcomes, but there was no difference in mean blood pressure between the control and intervention arms, suggesting the beneficial effect was not exclusively related to induced hypertension. One possibility is that the vasopressor reduced blood pressure variability, which preliminary data has shown to be detrimental after AIS, although that aspect of neurovascular coupling has not been adequately studied in the acute phase after AIS.

The reliance on IV vasopressors, which are only administered in the intensive care unit, is a fundamental limitation of prior research. An alternative, but untested, approach is to use the oral vasopressor midodrine hydrochloride. We hypothesize that frequent midodrine dosing after AIS can optimize collateral blood flow and help salvage the ischemic penumbra. The objective of this study is to develop tools to quantify midodrine's effect on blood pressure and the ischemic penumbra.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, ≥ 18 years old, with anterior circulation acute ischemic stroke on diffusion-weighted imaging (DWI) MRI, defined as predominant stroke burden in the frontal, parietal, or temporal lobes.
2. Demonstrable neurologic deficit due to stroke at randomization.
3. Within 12 hours of randomization, measured on CT or MR perfusion: a cerebral blood flow (CBF)/DWI ratio ≥1.25, an absolute difference between the CBF and DWI lesions of ≥15 mL, and a DWI volume between 20-100 mL. (Quantified with the Olea software)
4. Enrollment within 24 hours from stroke onset

Exclusion Criteria:

1. Endovascular therapy or intravenous tPA treatment for stroke
2. Acute myocardial infarction on ECG or troponin T >0.01 ng/mL.
3. History of cardiac disease, including myocardial infarction or unstable angina within the last 3 months, any history of clinically significant arrhythmia, symptomatic valvular disease, dilated cardiomyopathy, hypertrophic obstructive cardiomyopathy, left-ventricular assist device, or known ejection fraction < 25%.
4. Glomerular filtration rate < 50, serum creatinine >1.5 mg/dl, severe urinary retention, or end-stage renal disease on dialysis.
5. Coagulopathy, including INR >1.5, PTT >40, platelet count <75, or use of a novel anticoagulant in the last 3 days (e.g. dabigatran, rivaroxaban, apixaban).
6. Positive pregnancy test.
7. Clinical and laboratory evidence of thyrotoxicosis.
8. Severe Peripheral Vascular Disease or Raynaud's syndrome.
9. Systolic blood pressure (SBP) >180 or diastolic blood pressure (DBP) >100 immediately prior to randomization.
10. Allergy or history of adverse reaction to IV phenylephrine or midodrine.
11. Hemorrhage within the area of DWI lesion on MRI.
12. Indication for anticoagulation within 5 days of stroke onset.
13. Arterial dissection or cerebral aneurysm.
14. Pre-stroke modified Rankin score of >2.
15. Evidence of bacterial endocarditis.
16. Indication for carotid endarterectomy or stenting in next 5 days.
17. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.
18. Failure of post-stroke swallow evaluation and no alternative enteric access (e.g. nasogastric feeding tube, percutaneous endoscopic gastrostomy tube).
19. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study has been withdrawn
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Investigate the effect of midodrine on blood pressure mean and variability | During study drug administration

SECONDARY OUTCOMES:
The physiologic impact of midodrine. (daily mean flow velocity (MFV) in cm/second, of both the parent artery to the stroke and other reference intracranial arteries) | Days 1-4
  The outcome measure is a daily mean flow velocity (MFV) in cm/second, of both the parent artery to the stroke and other reference intracranial arteries.
The radiologic impact of midodrine. (percentage change in the size of the stroke (%) | Day 1 and Day 3-4
  The outcome measure is the size of the initial stroke in cm3 on day 1, and record the size of the final stroke in cm3 on the follow-up MRI at 3-4 days after enrollment. The investigators will then calculate a percentage change in the size of the stroke (%).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes